CLINICAL TRIAL: NCT00540761
Title: Natural History of Vulnerable Coronary Plaques
Brief Title: Identifying Vulnerable Plaques in Blood Vessels of the Heart Using a New Imaging Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2005-P000646; R01HL076398 (NIH)
Record Dates: First submitted 2007-09-24; First posted 2007-10-08 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Artery Disease; Atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- OFDI imaging (Experimental): OFDI catheter advanced to the distal coronary artery
  Interventions: Device: OFDI imaging
- Intravenous Ultrasound (Experimental): Randomization to determine whether Intravenous Ultrasound will be conducted before or after OFDI imaging.
  Interventions: Device: OFDI imaging

INTERVENTIONS:
Device: OFDI imaging — Intervention of OFDI system and Imaging of the culprit lesion using the OFDI system.

SUMMARY:
Atherosclerosis, a condition in which fatty deposits of plaque build up along the inner walls of arteries, is a condition that may increase the risk of having a heart attack. Previous studies have shown that the presence of a specific kind of plaque, known as vulnerable plaque, is often found in people who have had a heart attack. This study will use a new imaging technique called optical frequency domain imaging (OFDI) to examine the presence of vulnerable plaques in people with coronary artery disease.

DETAILED DESCRIPTION:
Atherosclerosis is a condition in which deposits of fat, cholesterol, and other substances build up along the inner walls of arteries; these deposits are known as plaque. As plaque builds up, it increases the risk of heart attack. Previous autopsy studies have shown that vulnerable plaques, a type of atherosclerotic plaque, are commonly found in people who have had a heart attack. Until recently it has been difficult to identify vulnerable plaques in people prior to their death. Many people who have coronary artery disease and are at risk of having a heart attack undergo angioplasty, a procedure that opens a narrowed or blocked blood vessel. During angioplasty, imaging devices are often used to take pictures of the inside of blood vessels. The most commonly used imaging device, an intravenous ultrasound (IVUS) catheter, is threaded through the blood vessels and uses sound waves to take pictures. An OFDI is a new type of catheter that takes more detailed pictures of blood vessel walls and plaques. The additional detail provided by OFDI images may improve detection of vulnerable plaques, which may help physicians identify people who are at high risk of having a heart attack. This study will use standard IVUS imaging and OFDI to examine vulnerable plaques within blood vessels of the heart and to evaluate any changes that occur over time in heart blood vessels and plaque.

This study will enroll participant with coronary artery disease who are undergoing angioplasty. At a baseline study visit, participants will first undergo an angiography procedure, in which x-ray pictures will be taken of the heart blood vessels. Participants will then be randomly assigned to undergo either the IVUS procedure followed by the OFDI procedure or vice versa. Repeat angiographies will occur after each imaging procedure. Next, participants will undergo angioplasty and a stent will be placed at the area of the blood vessel that is narrowed or blocked to keep the blood vessel open. Finally, participants will undergo repeat IVUS and OFDI procedures. For some participants, the study physician may perform the IVUS and OFDI procedures only after the angioplasty. Every six months and for a period of two years, participants will complete questionnaires about medication history and heart problems that may have occurred since the baseline visit.Blood collection will occur if this is done during office visit.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing PCTI for coronary artery disease
* Women with childbearing potential must have a negative pregnancy test within the 7 days prior to study entry

Exclusion Criteria:

* Kidney insufficiency (i.e., GFR<50ml/min)
* OR pregnancy
* OR participants who have had a ST elevation heart attack will be excluded for at least 72 hours post-heart attack and until cardiac enzymes return to normal. Participants who have had a non-ST elevation heart attack will be excluded if they have evidence of ongoing ischemia, defined as chest pain or new electrocardiogram (ECG) changes in the 12 hours prior to study entry and/or rising creatine kinase (CK) and CK-MB serum enzymes.
* OR high-risk and complex lesions, including tortuous blood vessels and lesions with thrombosis
* OR unprotected left main coronary artery disease
* OR enrolled in another investigational clinical trial within the 6 months prior to study entry
* OR severe peripheral vascular disease
* OR active ischemia
* OR congestive heart failure
* OR prior coronary artery bypass surgery
* OR emergent procedures
* OR inability to return for study follow-up procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Determine prevalence of vulnerable plaques | 2 years
  Number of subjects with vulnerable plaques

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Columbia Presbyterian Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waxman S, Freilich MI, Suter MJ, Shishkov M, Bilazarian S, Virmani R, Bouma BE, Tearney GJ. A case of lipid core plaque progression and rupture at the edge of a coronary stent: elucidating the mechanisms of drug-eluting stent failure. Circ Cardiovasc Interv. 2010 Apr;3(2):193-6. doi: 10.1161/CIRCINTERVENTIONS.109.917955. No abstract available. PMID 20407116